CLINICAL TRIAL: NCT01429454
Title: Randomized Double-Blind Trial of Omega 3 Fatty Acid Versus Placebo in Individuals at Risk for Psychosis
Brief Title: NAPLS Omega-3 Fatty Acid Versus Placebo Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kristin Cadenhead, M.D., Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAPLS- Omega3; U01MH081944 (NIH)
Record Dates: First submitted 2011-08-29; First posted 2011-09-07 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Psychosis
Keywords: Prodromal; Schizophrenia; Psychosis; Omega
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soybean-Corn Blend Capsule (Placebo Comparator): The placebo is a soybean/corn blend. Both the Omega-3FA and placebo are colored with carob (so shell is brown) and flavored with natural lemon-lime, to mask them.
  Interventions: Drug: Placebo
- Omega 3 long chain fatty acid (Experimental): The Omega-3 Fatty Acid compound will be manufactured by Ocean Nutrition Canada and contain an 2:1 proportion of EPA to DHA in which each capsule includes 370 mg EPA and 200 mg DHA as well as 2 mg/g Tocopherol. The dose will be two capsules per day for a total of 740 mg of EPA and 400 mg of DHA.
  Interventions: Drug: Omega-3 Long Chain Fatty Acid

INTERVENTIONS:
Drug: Omega-3 Long Chain Fatty Acid — : The Omega-3FA compound will be manufactured by Ocean Nutrition Canada and contain an 2:1 proportion of EPA to DHA in which each capsule includes 370 mg EPA and 200 mg DHA as well as 2 mg/g Tocopherol. The dose will be two capsules per day for a total of 740 mg of EPA and 400 mg of DHA.
  Other Names: Fish Oil, Ocean Nutrition
  Arms: Omega 3 long chain fatty acid
Drug: Placebo — The placebo is a soybean/corn blend. Both the Omega-3FA and placebo are colored with carob (so shell is brown) and flavored with natural lemon-lime, to mask them. The dose will be 2 capsules per day.
  Arms: Soybean-Corn Blend Capsule

SUMMARY:
The overall goal of the present study is to determine whether Omega-3 Fatty Acids potentially prevent onset of psychosis and improve clinical symptoms and functional outcome in youth and young adults at elevated clinical risk for schizophrenia and related disorders. The specific aims are: (1) To determine whether the rate of progression to psychosis is lower during six months of treatment with Omega-3 Fatty Acids compared to six months of treatment with placebo, (2) To determine whether Omega-3 Fatty Acids are more efficacious than placebo for prodromal symptoms, negative symptoms, and functioning, (3) To assess the safety and tolerability of Omega-3 Fatty Acids in this population, and (4) To conduct analyses of neuroimaging, neurocognitive, electrophysiological and other ancillary data to explore mechanistic explanations for the hypothesized benefits of Omega-3 Fatty Acids on clinical and functional outcomes (e.g., increases in white matter integrity and processing speed).

DETAILED DESCRIPTION:
Recruitment of subjects for clinical assessment and testing with dependent measures is considered for research purposes. Use will be made of existing data and records as the data obtained from this protocol will be used in combination with all data and records collected as part of the overall NAPLS study in which subjects are already enrolled. Individuals for this protocol will be recruited from UCSD's parent NAPLS study.

Experimental Treatment: This will be a 24-week, randomized, double-blind, placebo, fixed dose-controlled study designed to determine the acceptability and feasibility of Omega-3FA versus placebo in prodromal subjects assigned to treatments on a 1:1 basis. Omega-3FA will be administered as oral capsules given twice daily (BID). Ocean Nutrition Canada will prepare identical-looking Omega-3FA and placebo capsules. The investigators will include 128 prodromal subjects in the 6-month trial. All subjects will receive monthly clinical assessment. The study design and Omega-3FA formulation are designed to be compatible with that of another on-going trial conducted by investigators in Australia and Europe (the Neuropro Study sponsored by the Stanley Foundation), which would enable the data from the two studies to be combined for analysis on the primary (conversion) and most of the secondary and tertiary (symptoms, functioning) endpoints.

The proposed study will potentially further the development of novel treatment approach for the prodrome of psychosis. This research will provide empirical data regarding a lower risk, broad spectrum treatment, which could have important implications for public health as a pre-emptive intervention or treatment augmentation because of the potential to effect functional outcome. It is possible that subjects in the treatment group will show an improvement in symptoms. Study participants will receive extensive clinical evaluations and consultation from investigators with knowledge regarding psychosis.

The results of this study will increase the ability to provide alternative treatments with potentially fewer side effects for the prodrome of psychosis. The potential implication for primary and tertiary prevention of psychosis from these treatments is immeasurable. Through the development and utilization of strategies such as those proposed in this research the investigators could potentially discover the ability to delay the onset of psychosis and manage treatment more effectively with fewer side effects seen with traditional antipsychotic medication treatment. The importance of this to public health would be tremendous.

The use of Omega-3FA in an adolescent and young adult prodromal population is somewhat novel. Amminger et al 60 utilized a sample of 13 - 25 year old prodromal subjects to determine the potential benefit of EPA and DHA. Previous studies using Omega-3FA in adolescent and adult samples of psychotic subjects have produced no significant side effects. Some subjects reported a fishy aftertaste and mild gastrointestinal difficulties that dissipated with the discontinuation of Omega-3FA. Therefore the level of risk is considered minimal. This study offers subjects the possibility of direct benefit from participation because of the Omega-3FA and placebo treatments. It is also possible that the concurrent use of Omega-3FA will improve metabolic indices in all subjects. Because Omega-3FA is not specifically approved by the FDA for use in early psychosis, the investigators have received a certificate for an Investigational New Drug (IND) for the current Research Plan.

The sample of 128 prodromal subjects will be recruited from 8 sites over 16 months. UCSD is expected to recruit 14 of these prodromal subjects. The active treatment phase will be completed within 6 months, with 12-, 18-, and 24-month follow-ups. Each site will obtain institutional review board approval of the protocol. The UCLA site directed by Dr. Cannon and the UCSD site directed by Dr. Cadenhead, coordinate the trial, with responsibility for acquisition of the Omega-3 and placebo pills, group assignments, and data analysis.

Procedures

During the week prior to randomization and beginning study capsules, patients will undergo eligibility and baseline examinations. After beginning study capsules, patients will be scheduled for 6 monthly follow-up visits as well as 12-, 18-, and 24-month follow-ups.

Omega-3FA and Placebo: The Omega-3FA compound will be manufactured by Ocean Nutrition Canada and contain an 2:1 proportion of EPA to DHA in which each capsule includes 370 mg EPA and 200 mg DHA as well as 2 mg/g Tocopherol. The dose will be two capsules per day for a total of 740 mg of EPA and 400 mg of DHA. The ratio and dose of Omega-3FA were selected based on previous data from controlled trials that demonstrates the efficacy of EPA in trials with schizophrenia patients37, 38 and the potential benefit of a low dose of DHA in combination with EPA per the Amminger study60 in prodromal patients. The placebo is a soybean/corn blend. Both the Omega-3FA and placebo are colored with carob (so shell is brown) and flavored with natural lemon-lime, to mask them. Certificates of analysis for the Omega-3FA and placebo compounds are included in the Appendix. Ongoing testing by independent laboratories will assure the levels of Omega-3FA in capsules, stability, and absence of any contaminants, including toxic substances in this product. Stability and toxicology testing will be provided by Siliker Canada Co. UCLA will receive the compounds and assign coded numbers to packets before distribution to sites and thereby administer the double blind design.

Antipsychotics: Prodromal subjects currently on anti-psychotic medication will be excluded from the study. It is possible that prodromal subjects will develop worsening symptoms and require such treatments during the course of the trial, which is allowed. All concomitant treatment will be recorded.

Antidepressants: Prodromal patients currently on anti-depressant medication will be included in the study; randomization to Omega-3FA vs. placebo will be stratified on anti-depressant medication status.

Background Diet: Baseline diet characterization will be assessed using a systematic checklist. The investigators considered using an open-ended diary that requires recording of all food intake, but it seems unlikely that adolescents with early psychosis symptoms would comply to a satisfactory degree. The checklist is easy to complete and is more likely to be accurate than unstructured self-reports. The list includes foods that are rich in Omega-3FA. It will be given to the family at the first screening visit, and will be collected for the two consecutive weeks preceding entry into the treatment phase. Intake will be categorized as low (0-1 serving/wk of Omega-3FA rich diet), intermediate (2-3 servings/wk), or high (4 or more servings/wk). In addition fasting erythrocyte FA composition will be assessed to use as another means of controlling for background diet at baseline.

Laboratory and Metabolic Measures: After confirming eligibility for the study, a urine sample will be taken for a drug screen, and a serum pregnancy test on females. Fasting erythrocyte FA composition will be quantified at baseline, month 3 and month 6 using capillary gas chromatography. The ratio of Omega-6 to 3FAs will be used to index pretreatment vs posttreatment FA composition as an objective measure of treatment adherence, to assess for dietary differences between subjects and assure that subjects on placebo are not taking Omega-3FA supplementation from an outside source. Thiobarbituric Acid Reactive Substances (TBARS) will be used for screening and monitoring lipid peroxidation before and after the treatment trial. In addition, to assess metabolic parameters, baseline measures of fasting glucose and lipids, weight, abdominal girth and blood pressure will be obtained and repeated at the end of the trial.

Other Concomitant Medications: Subjects may continue doses of antidepressant, mood stabilizer, or stimulant medication as prescribed independently of their participation in this trial. Antipsychotic mediation will not be permitted unless subjects develop worsening symptoms and require antipsychotic medication during the course of the trial. All concomitant treatment will be recorded.

Concomitant Psychotherapy: During the 6-month active treatment phase, all subjects will be receive up to 6 sessions of supportive case management, as needed, as part of their evaluations by psychological staff. Staff members will provide support and address the young person's efforts to cope with symptoms and functional deficits. In addition, subjects will be permitted to participate in any outside of study supportive psychotherapy, with all concomitant psychological treatments recorded.

Study Management: Prior to study launch, study investigators and other key personnel will participate in several conference calls to provide training on study procedures, including recruitment strategies, inclusion and exclusion criteria, use of rating scales, and data management procedures.

After study launch, the co-PIs at the UCLA and UCSD sites will chair conference calls every two weeks attended by each site PI and study coordinator. Reports on enrollment and data completeness will be discussed regularly, along with issues brought up by sites.

Data Management: UCLA will provide the central data management site for the proposed study, and the University of Calgary site (Dr. Addington) will be responsible for overall NAPLS data management. This will be done through a centralized Oracle database with web based data input that will facilitate study coordination, data checks and early identification of faulty procedures and data errors. The database is secure, robust and easy for clinical investigators and staff to learn and use. Security access can be limited to site level with a range of access for different levels of personnel. Data entry will be of the highest standards such that each data element/field is defined with ranges, allowed values and size.

Post-treatment Biomarkers Assessment

Patients enrolled in this trial will be participants in the parent study "Predictors and Mechanisms of Conversion to Psychosis." In the context of that study, participants are assessed with MRI/DTI, electrophysiology (including PPI), neuropsychological testing at baseline and 12- and 24-month follow-ups. Given that participants in the Omega-3FA study will complete the active treatment phase at 6 months, it is desirable to add an additional biomarkers assessment point for those subjects at the 6-month (end of treatment) follow-up.

Assessments

Sources of material will come primarily from the participant, in the form of the results of questionnaires, clinical interviews, physical exam, and blood draws. All participants will undergo a series of clinical, functional, neurocognitive, neuroimaging and electrophysiological assessments, which are part of the overall NAPLS study, before and after the 6 months of Omega-3FA versus placebo. Therefore data collected as part of the parent study will be assessed for changes that may be attributable to these treatment trials. Biological specimens (blood) will be collected at baseline, 3 months and 6 months of the Omega-3FA trial to help evaluate the level of Omega-3FA in the diet and metabolic indices as well (urine) to evaluate substance use at time of testing.

For minors, a parent/legal guardian may provide additional information useful for clinical or historical data. Written and oral consent will be obtained from participants, or their legal guardian for minor participants. Assent will be obtained from minors. Only study personnel directly associated with the research will have access to individually identifiable information.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included if they are treatment-seeking patients between the ages of 12 and 30 who meet diagnostic criteria for a possible prodromal syndrome and are part of the ongoing NAPLS study.

Exclusion Criteria:

* use of antipsychotic medication in the previous month.
* concomitant medical or neurological illness.
* history of significant head injury.
* alcohol or drug abuse (excluding nicotine) in the past month or dependence in the past three months.
* screening full scale estimated IQ < 80.
* active suicidal or homicidal ideation.
* pregnancy or lactation.
* allergies to seafood or seafood related products or no history of seafood consumption

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 127 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin S Cadenhead, MD, Principal Investigator — UCSD
Locations (9):
- United States (8):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Harvard, Boston, Massachusetts
  - Zucker Hillside Hospital, Glen Oaks, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
- University of Calgary, Calgary, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Soybean-Corn Blend Capsule | Omega 3 Long Chain Fatty Acid
Started | 62 | 65
Completed | 35 | 35
Not Completed | 27 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Soybean-Corn Blend Capsule | Omega 3 Long Chain Fatty Acid | Total
Number analyzed (Participants) | 62 | 65 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 30 | 62
  Between 18 and 65 years | 30 | 35 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.37 (4.66) | 18.95 (4.65) | 18.69 (4.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 33 | 38 | 71
Region of Enrollment [Number; unit: participants]
  Canada | 13 | 14 | 27
  United States | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Rate of Conversion to Psychosis.
Description: The rate of conversion to psychosis among prodromal patients assigned at random to Omega-3 Fatty Acids at 12 months will be significantly lower than that among patients assigned to placebo.The Structured Interview for Prodromal Syndromes (SIPS) include the "Presence of Psychotic Syndrome (POPS)" scale that determines if the criteria for conversion to psychosis are met. The scale is binary, a 1 equals conversion and 0 equals non-conversion.
Time Frame: 12 months
Population: The population included participants who met the criteria for Clinical High Risk for Psychosis
Measure: Count of Participants; unit: Participants
Groups:
- Omega 3 Fatty Acid: Omega 3 Fatty Acid Supplementation
- Placebo: Soybean/corn blend
Arm/Group | Omega 3 Fatty Acid | Placebo
Number analyzed (Participants) | 65 | 62
Participants | 4 | 3
Statistical Analysis 1: Comparison: Omega 3 Fatty Acid vs Placebo; Test type: Superiority; p = .51, Chi-squared; Cox Proportional Hazard = .36

2. Secondary Outcome: Scale of Prodromal Symptoms (SOPS) Total Score (Indexing Severity of Positive, Negative, and General Symptoms)
Description: The reduction from baseline in the Scale of Prodromal Symptoms (SOPS) total score (indexing severity of positive, negative, and general symptoms) at 6 and 12 months will be significantly greater in prodromal patients assigned at random to Omega-3 Fatty Acids than in patients assigned to placebo.
  Minimum SOPS score= 0 Maximum SOPS score= 114
  Higher Total SOPS score does not necessarily mean the subject is more "psychotic" as the aggregate score is that of four independent categorically defined symptom subscales, including: Positive Symptoms Scale, Negative Symptoms Scale, Disorganized Symptoms Scale, and General Symptoms Scale. However, a higher Total SOPS score would likely indicate an individual is presenting with more overall symptoms.The Structured Interview for Prodromal Syndromes (SIPS) determines if the criteria for conversion to psychosis has been met.
Time Frame: 6 month follow up
Population: These subject numbers represent the number of participants who completed the 6 month evaluation and had symptom ratings performed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Soybean-Corn Blend Capsule
Arm/Group | Omega 3 Fatty Acid | Placebo
Number analyzed (Participants) | 34 | 36
score on a scale | 27.2 (12.4) | 28.8 (15.4)
Statistical Analysis 1: Comparison: Omega 3 Fatty Acid vs Placebo; Test type: Superiority; p > 0.10, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Soybean-Corn Blend Capsule | Omega 3 Long Chain Fatty Acid
Serious Adverse Events (participants affected / at risk) | 4/62 | 2/65
Other Adverse Events (participants affected / at risk) | 48/62 | 53/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soybean-Corn Blend Capsule (N=62) | Omega 3 Long Chain Fatty Acid (N=65)
Hospitalization due to suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Hospitalization due to severe stomach pain diagnosed as Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Attempted suicide (Psychiatric disorders) | 1 (1) | 0 (0) — Overdose of pills
Attempt to quiet auditory hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) — With excess Quetiapine ingestion
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Evaluated at the Emergency Department
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soybean-Corn Blend Capsule (N=62) | Omega 3 Long Chain Fatty Acid (N=65)
Sedation/drowsiness (Nervous system disorders) | 28 (28) | 36 (36)
Irritability (General disorders) | 36 (36) | 33 (33)
Headache (General disorders) | 32 (32) | 31 (31)
Insomnia (General disorders) | 26 (26) | 35 (35)
Sleep disturbance, other (General disorders) | 26 (26) | 35 (35)
Fatigue/weakness (General disorders) | 27 (27) | 31 (31)
Excitement/nervousness (General disorders) | 26 (26) | 29 (29)
Appetite decrease (General disorders) | 25 (25) | 28 (28)
Memory problems (General disorders) | 25 (25) | 25 (25)
Sensory perception abnormality (General disorders) | 24 (24) | 26 (26)
Malaise (General disorders) | 21 (21) | 25 (25)
Stomach/abdominal discomfort (Gastrointestinal disorders) | 22 (22) | 24 (24)
Hallucinations (Psychiatric disorders) | 23 (23) | 20 (20)
Nasal congestion (General disorders) | 19 (19) | 24 (24)
Mentation impaired (General disorders) | 19 (19) | 21 (21)
Dizziness/faintness (General disorders) | 14 (14) | 24 (24)
Nausea/vomiting (Gastrointestinal disorders) | 19 (19) | 19 (19)
Appetite increase (General disorders) | 19 (19) | 19 (19)
Weight gain (Gastrointestinal disorders) | 17 (17) | 21 (21)
Tinnitus/difficulty hearing (Ear and labyrinth disorders) | 19 (19) | 17 (17)
Dry mouth (General disorders) | 15 (15) | 21 (21)
Weight loss (Gastrointestinal disorders) | 14 (14) | 20 (20)
Muscle twitching (General disorders) | 18 (18) | 15 (15)
Depersonalization (Psychiatric disorders) | 16 (16) | 16 (16)
Muscle cramps (General disorders) | 14 (14) | 18 (18)
Tachycardia/palpitations (Cardiac disorders) | 17 (17) | 15 (15)
Derealization (Psychiatric disorders) | 15 (15) | 15 (15)
Ataxia/impaired coordination (Musculoskeletal and connective tissue disorders) | 13 (13) | 17 (17)
Chest pain (Cardiac disorders) | 12 (12) | 17 (17)
Delusions (Psychiatric disorders) | 13 (13) | 15 (15)
Sweating excessively (General disorders) | 10 (10) | 17 (17)
Vision blurred (Eye disorders) | 12 (12) | 14 (14)
Tremor (General disorders) | 15 (15) | 11 (11)
Speech slurred (General disorders) | 14 (14) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 14 (14) | 10 (10)
Dermatitis/allergy (General disorders) | 14 (14) | 10 (10)
Other (General disorders) | 6 (6) | 17 (17)
Libido decrease (General disorders) | 8 (8) | 11 (11)
Salivation increase (General disorders) | 7 (7) | 10 (10)
Constipation (Gastrointestinal disorders) | 5 (5) | 11 (11)
Abnormal muscle tone/movement (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8)
Hyperventilation (General disorders) | 6 (6) | 8 (8)
Libido increase (General disorders) | 6 (6) | 8 (8)
Edema (General disorders) | 5 (5) | 4 (4)
Urination problems (Renal and urinary disorders) | 0 (0) | 3 (3)
Fishy burp (General disorders) | 6 (6) | 10 (10)

LIMITATIONS AND CAVEATS:
The high rate of attrition was a limitation in being able to fully assess the psychotic conversion outcome of this study or outcome greater than 6 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT01429454/Prot_SAP_000.pdf